CLINICAL TRIAL: NCT06094920
Title: Optimization of Albuminuria-Lowering Therapies for Individual Patients With Type 2 Diabetes Using Empagliflozin and Finerenone in a Pilot Remote Clinical Trial.
Brief Title: Treatment Optimization for Patients With Type 2 Diabetes Using Empagliflozin and Finerenone in a Remote Clinical Trial
Acronym: Optimize@Home
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18253
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus Type 2 With Proteinuria; Diabetes Mellitus, Type 2; Diabetes Mellitus; Diabetes; Diabetes Complications; Albuminuria; Chronic Kidney Diseases; Chronic Kidney Disease Due to Type 2 Diabetes Mellitus; Chronic Kidney Disease stage3; Chronic Kidney Disease stage4; CKD; CKD Stage 3; CKD Stage 4
Keywords: Type 2 diabetes; Diabetes Mellitus, Type 2; Albuminuria; Diabetes Mellitus; Diabetes Mellitus Type 2 with Proteinuria; Personalized Medicine; Decentralized; Remote clinical trial; Remote data collection; Individualized; Treatment optimalization; CKD; Chronic Kidney Disease; Albuminuria-Lowering Therapies; Empagliflozin; Finerenone; SGLT2 inhibitors; MRA; Sodium Glucose Co-Transporter 2; Mineralocorticoid Receptor Antagonist
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Diabetes Complications; Albuminuria; Renal Insufficiency, Chronic | interventions — empagliflozin; finerenone; Digital Technology

STUDY DESIGN:
Intervention Model Description: Eligible participants will be assigned to a 3-week treatment period with the SGLT2 inhibitor empagliflozin 10 mg/day, in accordance with guidelines. After 2 weeks, albuminuria levels will be assessed to determine the individual albuminuria response. Depending on the response (decrease or increase), participants will be allocated to one of three treatment regimens following the 3-week empagliflozin treatment period:
  A. Albuminuria reduction >30% and the remaining albuminuria level is <30 mg/g: continue empagliflozin for an additional four weeks.
  B. Albuminuria reduction >30% or >0 and ≤30%, and the remaining albuminuria level is >30 mg/g: continue empagliflozin for an additional four weeks and intensify treatment by adding finerenone for four weeks.
  C. No albuminuria reduction or increase: discontinue empagliflozin and switch to finerenone for four weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- A. Good albuminuria response after 2 weeks empagliflozin 10 mg/day (Other): Albuminuria reduction >30% and the remaining albuminuria level is <30 mg/g: continue empagliflozin 10 mg/day for an additional four weeks.
  Interventions: Drug: Empagliflozin 10 MG; Device: Withings BPM Connect; Device: Withings Body; Diagnostic Test: PeeSpot Urine Collection Device; Diagnostic Test: Hem-Col Capillary Blood Collection Device; Behavioral: Questionnaire: participants' perspectives toward the feasibility of participation in a trial at home with digital technologies
- B. Moderate albuminuria response after 2 weeks empagliflozin 10 mg/day (Other): Albuminuria reduction >30% or >0 and ≤30%, and the remaining albuminuria level is >30 mg/g: continue empagliflozin 10 mg/day for an additional four weeks and intensify treatment by adding finerenone 10 or 20 mg/day for four weeks (dosage depends on eGFR levels).
  Interventions: Drug: Empagliflozin 10 MG; Drug: Finerenone; Device: Withings BPM Connect; Device: Withings Body; Diagnostic Test: PeeSpot Urine Collection Device; Diagnostic Test: Hem-Col Capillary Blood Collection Device; Behavioral: Questionnaire: participants' perspectives toward the feasibility of participation in a trial at home with digital technologies
- C. No albuminuria reduction after 2 weeks empagliflozin 10 mg/day (Other): No albuminuria reduction or increase: discontinue empagliflozin and switch to finerenone 10 or 20 mg/day for four weeks (dosage depends on eGFR levels).
  Interventions: Drug: Finerenone; Device: Withings BPM Connect; Device: Withings Body; Diagnostic Test: PeeSpot Urine Collection Device; Diagnostic Test: Hem-Col Capillary Blood Collection Device; Behavioral: Questionnaire: participants' perspectives toward the feasibility of participation in a trial at home with digital technologies

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Oral administration
  Other Names: Jardiance; A10BK03; (2S,3R,4R,5S,6R)-2-[4-chloro-3-[[4-[(3S)-oxolan-3-yl]oxyphenyl]methyl]phenyl]-6-(hydroxymethyl)oxane-3,4,5-triol
  Arms: A. Good albuminuria response after 2 weeks empagliflozin 10 mg/day; B. Moderate albuminuria response after 2 weeks empagliflozin 10 mg/day
Drug: Finerenone — Oral administration.
  Finerenone treatment may be initiated if serum potassium levels are ≤5.0 mmol/L. Conversely, if serum potassium levels are >5.0 mmol/L, the initiation of finerenone treatment should be avoided. In such cases, a second serum potassium measurement will be performed two days later. If serum potassium levels are ≤5.0 mmol/L, these patients can still be considered for inclusion. However, if serum potassium levels are >5.0 mmol/L again, these patients will be excluded, and an assessment of the underlying cause(s) of hyperkalaemia will be conducted.
  The recommended initial dose of finerenone is determined based on eGFR, which will be assessed prior to the commencement of the trial. If eGFR is ≥60 mL/min/1.73m2, the dose will be set at 20 mg once daily. If eGFR is ≥25 to <60, the dose will be set at 10 mg once daily. Participants with an eGFR <25 are not advised to undergo finerenone treatment and will be excluded from the study.
  Other Names: Kerendia; C03DA05; (4S)-4-(4-cyano-2-methoxyphenyl)-5-ethoxy-2,8-dimethyl-1,4-dihydro-1,6-naphthyridine-3-carboxamide
  Arms: B. Moderate albuminuria response after 2 weeks empagliflozin 10 mg/day; C. No albuminuria reduction after 2 weeks empagliflozin 10 mg/day
Device: Withings BPM Connect — CE marked and clinically validated blood pressure monitor. Clinical trial results are within the margin of acceptance defined by the internationally recognized evaluation standard of blood pressure monitors ANSI/AAMI/ISO 81060-2:2013, EN ISO 81060-2:2014, developed by the European Society of Hypertension, British Hypertension Society and Association for the Advancement of Medical Instrumentation/American Heart Association.
  Blood pressure will be measured by the participants once daily on 40 days. Three consecutive measurements are taken.
Device: Withings Body — CE marked and clinically validated advanced Wi-Fi smart scale.
  Body weight will be measured by the participants once daily on 49 days.
Diagnostic Test: PeeSpot Urine Collection Device — Biochemical urine data will be collected using first-morning void urine samples. Participants will obtain urine samples with the PeeSpot device, a validated tool designed for the collection and preservation of small urine volumes. This device comprises a urine absorption pad, a holder, a tube, and a lid. Patients can void directly onto the absorption pad while it is placed in the holder. Following voiding, the pad and holder are inserted into the tube, sealed with the lid, and stored in a refrigerator until they are sent to the laboratory using a biological materials envelope (PolyMed, DaklaPack, Europe). Through the incorporation of an inert hygroscopic polymer, the pad efficiently absorbs 1.2 mL of urine, and with the addition of various preservatives, the urine remains stable for up to four days. The investigators will employ the PeeSpot to determine the first-morning void levels of albumin, creatinine, sodium, potassium, glucose, urea, and osmolality once daily on 28 days.
Diagnostic Test: Hem-Col Capillary Blood Collection Device — Capillary blood samples will be obtained using a BD Microtainer® Contact-Activated Lancet (Franklin Lakes, New Jersey, USA) once daily on 17 days. These blood samples will be collected into Hem-Col® tubes (Hem-Col, Labonovum, Limmen, the Netherlands), specifically designed for collection of capillary blood acquired through a finger prick. The Hem-Col microtube is equipped with an anticoagulant and a preservation buffer, enhancing the stability of analytes in whole blood. These Hem-Col tubes have the dimensions of standard blood collection tubes and are constructed from polyethylene, featuring a pierceable cap made of thermoplastic elastomers. Each tube incorporates a liquid barrier, with the inner part preventing the loss of Hem-Col preservation fluid and the outer part serving as a scoop for collecting blood from a finger prick. The Hem-Col lithium heparin tubes will be utilized for the analysis of creatinine, potassium, hsCRP, haematocrit, cystatin C, and fasting plasma glucose.
Behavioral: Questionnaire: participants' perspectives toward the feasibility of participation in a trial at home with digital technologies — Participant perspectives regarding the feasibility of participating in a home-based trial will be evaluated using a digital questionnaire. This questionnaire includes inquiries adapted from the validated Telehealth Usability Questionnaire, supplemented with additional questions employed in prior studies that assessed the feasibility of decentralized clinical trials. The web application Research Electronic Data Capture 10.0.23 (REDCap - www.projectredcap.org) will facilitate the administration of these digital questionnaires. Participants will receive a link to access the digital questionnaires via email. Weekly telephone calls will be conducted to evaluate adherence to study procedures and monitor the occurrence of adverse events.

SUMMARY:
The goal of this clinical trial is to determine the feasibility of remote clinical trial conduct in patients with type 2 diabetes and elevated albuminuria. The main questions it aims to answer are:

* What is the feasibility (and advantages) of remote clinical trial conduct with multiple medications in patients with type 2 diabetes and elevated albuminuria?
* What is the individual response to the SGLT2 inhibitor empagliflozin in urine albumin-creatinine ratio?
* What is the individual response to the SGLT2 inhibitor empagliflozin in systolic blood pressure, body weight, eGFR, and fasting plasma glucose?
* Can suboptimal treatment responses to empagliflozin be overcome by the addition or substitution with finerenone?

Participants will collect all study data in the comfort of their own environments

* First-morning void urine samples
* Capillary blood samples
* Blood pressure
* Body weight

Participants will be assigned to a 3-week treatment period with empagliflozin 10 mg/day. Based on the albuminuria response after 2 weeks, participants will be allocated to one of three treatment regimens after the 3-week treatment period with empagliflozin:

* Continue empagliflozin for 4 more weeks (good response).
* Continue empagliflozin for 4 more weeks and add finerenone 10 or 20 mg will be added for 4 weeks (moderate response).
* Stop empagliflozin and start finerenone 10 or 20 mg for 4 weeks (no response)

DETAILED DESCRIPTION:
Rationale:

The treatment of cardiovascular and kidney-related complications associated with type 2 diabetes has made significant progress in recent years. Clinical trials have demonstrated the clinical benefits of sodium glucose co-transporter 2 (SGLT2) inhibitors and the selective non-steroidal mineralocorticoid receptor antagonist (MRA) finerenone. Guidelines from professional nephrology and cardiology associations now recommend the use of SGLT2 inhibitors and finerenone for all patients with type 2 diabetes and chronic kidney disease (CKD). Although guidelines recommend the use of these new drug classes for all patients, the adoption in clinical practice has been slow, with implementation barriers existing at the healthcare facility, physician, and patient levels.

Despite the beneficial effects of these new drug classes on a population level, resulting in a reduction in the relative risks of cardiovascular and kidney outcomes, a high residual risk remains, which is closely associated with high levels of albuminuria. This remaining risk can, in part, be attributed to sub-optimal individual responses to SGLT2 inhibitors and finerenone. The investigators' previous research has demonstrated substantial variability in individual albuminuria responses to SGLT2 inhibitors and MRAs among patients, indicating that some patients benefit from SGLT2 inhibitors, others from finerenone, and yet another group requires a combination of both agents for optimal cardiovascular and kidney protection.

To leverage technological advancements and evaluate drug efficacy and safety at an individual patient level, the investigators propose a pilot remote (home-based) clinical trial aimed at demonstrating the feasibility and advantages of conducting a remote clinical trial involving multiple medications to identify optimal therapy with the least pill burden for each patient. This trial will also assess patient experiences with data collection conducted remotely. This would potentially help (1) to facilitate the implementation of guideline-recommended treatments, (2) to optimize the guideline-recommended treatments for each individual, and (3) to evaluate individual drug responses and tailor therapy to each patient. Ultimately, the investigators' goal is to transition patient care from clinical settings (hospitals or general practitioner practices) to the home environment, making treatment regimen adjustments based on remotely collected data. This shift aims to minimize patient visits and enhance patient participation in optimizing their therapy in line with established guidelines.

Objective:

The primary objective is to determine the feasibility and advantages of remote clinical trial conduct with multiple medications in patients with type 2 diabetes and elevated albuminuria.

The secondary objectives are to:

* Determine the individual response to the SGLT2 inhibitor empagliflozin in urine albumin-creatinine ratio (UACR).
* Determine the individual response to the SGLT2 inhibitor empagliflozin in systolic blood pressure, body weight, estimated glomerular filtration rate (eGFR), and fasting plasma glucose.
* Assess if suboptimal treatment responses to empagliflozin can be overcome by the addition or substitution with finerenone.

Main trial endpoints:

The main trial endpoints are:

* Questionnaire results: participants' perspectives toward the feasibility of participation in a trial at home with digital technologies.
* Number and percentage of urine collections not received at the laboratory or unable to be analysed.
* Number and percentage of missed blood pressure or body weight measurements.
* Treatment adherence: pill count and medication concentration in urine samples.

Secondary trial endpoints:

The secondary trial endpoints are:

* Change from baseline in UACR from start to end of treatment with empagliflozin.
* Change from baseline in systolic blood pressure, body weight, eGFR, and fasting plasma glucose from start to end of treatment with empagliflozin.
* (Additive) treatment effects on UACR, systolic blood pressure, body weight, eGFR, and fasting plasma glucose from start to end of treatment after the addition or substitution with finerenone.

Trial design:

This is a single-centre, prospective, open-label, decentralised, crossover pilot study where participants are participating for 10 weeks.

Trial population:

Adult participants with type 2 diabetes, UACR >4.5 mg/mmol (>40 mg/g) and ≤300 mg/mmol (≤2655 mg/g), and eGFR ≥25 mL/min/1.73m2 who are on stable treatment with an angiotensin-converting enzyme (ACE) inhibitor or angiotensin II receptor blocker (ARB), unless not tolerated. The investigators aim to recruit 10 participants who are receiving care in primary or secondary healthcare settings.

Interventions:

Eligible participants will be assigned to a 3-week treatment period with the SGLT2 inhibitor empagliflozin 10 mg/day, in accordance with guidelines. After 2 weeks, albuminuria levels will be assessed to determine the individual albuminuria response. Depending on the response (decrease or increase), participants will be allocated to one of three treatment regimens following the 3-week empagliflozin treatment period:

A. Albuminuria reduction >30% and the remaining albuminuria level is <30 mg/g: continue empagliflozin 10 mg/day for an additional four weeks.

B. Albuminuria reduction >30% or >0 and ≤30%, and the remaining albuminuria level is >30 mg/g: continue empagliflozin 10 mg/day for an additional four weeks and intensify treatment by adding finerenone 10 or 20 mg/day for four weeks (dosage depends on eGFR levels).

C. No albuminuria reduction or increase: discontinue empagliflozin and switch to finerenone 10 or 20 mg/day for four weeks (dosage depends on eGFR levels).

Ethical considerations relating to the clinical trial including the expected benefit to the individual participants or group of patients represented by the trial participants as well as the nature and extent of burden and risks:

Both medicinal products are indicated for the treatment of patients with type 2 diabetes supported by multiple large-scale international clinical trials. Empagliflozin is currently marketed and recommended for adult patients with CKD, both with and without diabetes. It can be prescribed to individuals with an eGFR as low as 20 mL/min/1.73m2. The efficacy and safety of empagliflozin have been demonstrated in numerous parallel randomised controlled trials involving over 25,000 patients with type 2 diabetes. The most frequently reported adverse reaction when used in conjunction with sulfonylureas or insulin was hypoglycaemia. Other commonly reported adverse reactions included volume depletion, urinary tract infections, genital infections, thirst, constipation, (generalised) pruritus, rash, increased urination, and elevated serum lipids. Finerenone is currently marketed and recommended for use in adult patients with type 2 diabetes and stage 3 or 4 CKD, as indicated by an eGFR <60 mL/min/1.73m2 and a UACR >3 mg/mmol. The efficacy and safety of finerenone have been established through multiple parallel randomised controlled trials involving more than 10,000 patients with CKD and type 2 diabetes. The most frequently reported adverse reactions during treatment with finerenone was hyperkalaemia (14.0%). Other common adverse reactions included hyponatremia, hyperuricemia, hypotension, pruritus, and decreased GFR. Due to the modest increase in risk of hyperkalaemia with finerenone, the investigators will include only patients with serum potassium <5.0 mmol/L in this study. Guidelines from professional nephrology and cardiology associations now recommend the use of SGLT2 inhibitors and finerenone for all patients with type 2 diabetes and CKD. Participants who exhibit a favourable response to empagliflozin and/or finerenone and whose characteristics align with the criteria for clinical use can consult their treating physician to evaluate the ongoing use of empagliflozin and/or finerenone and to determine if additional laboratory assessments are necessary. Participating patients will be given free study medications and an opportunity to identify the optimal personalised regimen evaluated by objective assessment under the supervision of the study team.

Participants visit the study site on three occasions: a screening visit, baseline visit, and an end-of-study visit. This trial will adopt a decentralised approach in which participants will measure and collect study variables at home, including biochemical urine and capillary blood data, blood pressure, and body weight. This will minimize patient travel, study site visits, and facilitate clinical trial participation. Instructions for remote data collection are provided during the second study visit, and data collection occurs on scheduled days.

Biochemical urine data are obtained from first-morning void urine samples using the PeeSpot device. Capillary blood samples are collected using a BD Microtainer Contact-Activated lancet and Hem-Col tubes. Participants send their urine and capillary blood samples to the laboratory by mail. To familiarize participants with blood collection procedures, they perform a capillary blood sample collection at the study site during the second visit under the supervision of a trained lab technician. Additionally, a venous blood sample is drawn during the second study visit to enable comparison of clinical chemistry assessments between capillary and venous blood samples. Blood pressure and body weight measurements are performed using validated smart devices. Blood pressure and body weight measurements will be automatically stored in the corresponding mobile application.

The overall study duration is expected to be 10 weeks. The expected time commitment for participants is approximately 25 hours, including at-home measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of type 2 diabetes
* UACR >4.5 mg/mmol (>40 mg/g) and ≤300 mg/mmol (≤2655 mg/g)
* eGFR ≥25 mL/min/1.73m2
* On a stable dose of an ACE inhibitor/ARB if tolerated
* Willing to sign informed consent.
* Proficiency in the Dutch language

Exclusion Criteria:

* Diagnosis of type 1 diabetes
* Already treated with any SGLT2 inhibitor or MRA
* Unable to monitor blood pressure or body weight or handle digital technologies.
* Heart failure New York Heart Association (NYHA) Class II to IV requiring MRA treatment
* Acute coronary syndrome event within 6 months
* Serum potassium >5 mmol/L repeat value after repeated measurement
* Evidence of severe hepatic impairment determined by any of one: ALT or AST values exceeding 3 times ULN, a history of hepatic encephalopathy, a history of oesophageal varices, or a history of portocaval shunt.
* Active pregnancy or breastfeeding
* History of kidney or liver transplant
* Unstable or rapidly progressing renal disease.
* Active malignancy
* Suggestive evidence of adrenal insufficiency
* History of severe hypersensitivity or contraindications to any SGLT2 inhibitor or MRA
* Uncontrolled arterial hypertension (mean sitting systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg)
* Any medication, surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of medications including, but not limited to any of the following:
* History of active inflammatory bowel disease within the last 6 months
* Major gastrointestinal tract surgery as decided by the physician.
* Pancreatitis within the last 6 months
* Gastrointestinal ulcers and/or bleeding within the last 6 months
* Evidence of urinary obstruction or difficulty in voiding at screening
* Participation in any clinical trial within 3 months prior to initial dosing
* Donation or loss of ≥400 mL of blood within 8 weeks prior to initial dosing
* Confirmed lactose intolerance demonstrated with a lactose intolerance test.
* History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during screening or according to investigator's assessment.
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol.
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
* Women of childbearing potential (WOCBP):
* WOCBP who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of the study drug in such a manner the risk of pregnancy is minimised.
* WOCBP must have a negative serum or urine pregnancy test result (minimum sensitivity 25 IU/L or equivalent of HCG) at screening.

WOCBP comprises women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who are not post-menopausal (see definition below). The following women are NOT considered as WOCBP:

* Women using the following methods to prevent pregnancy: oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as intrauterine devices or barrier methods (diaphragm, condoms, spermicides).
* Women who are practicing abstinence.
* Women who have a partner who is sterile (e.g. due to vasectomy).

Post-menopause is defined as:

* Women who have had amenorrhea for >12 consecutive months (without another cause) and who have a documented serum follicle-stimulating hormone (FSH) level >35 mIU/mL.
* Women who have irregular menstrual periods and a documented serum FSH level >35 mIU/mL.
* Women who are taking hormone replacement therapy (HRT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Questionnaire results | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  Participants' perspectives toward the feasibility of participation in a trial at home with digital technologies
Remote urine collection | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  Number and percentage of urine collections not received at the laboratory or unable to be analysed
Remote blood pressure measurements | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  Number and percentage of missed blood pressure measurements
Remote body weight measurements | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  Number and percentage of missed body weight measurements
Treatment adherence | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  Pill count and medication concentration in urine samples

SECONDARY OUTCOMES:
Individual UACR response to empagliflozin | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  Change from baseline in UACR from start to end of treatment with empagliflozin.
Individual systolic blood pressure response to empagliflozin | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  Change from baseline in systolic blood pressure from start to end of treatment with empagliflozin.
Individual body weight response to empagliflozin | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  Change from baseline in body weight from start to end of treatment with empagliflozin.
Individual eGFR response to empagliflozin | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  Change from baseline in eGFR from start to end of treatment with empagliflozin.
Individual fasting plasma glucose response to empagliflozin | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  Change from baseline in fasting plasma glucose from start to end of treatment with empagliflozin.
(Additive) treatment effects finerenone on UACR | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  (Additive) treatment effects on UACR from start to end of treatment after the addition or substitution with finerenone.
(Additive) treatment effects finerenone on systolic blood pressure | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  (Additive) treatment effects on systolic blood pressure from start to end of treatment after the addition or substitution with finerenone.
(Additive) treatment effects finerenone on body weight | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  (Additive) treatment effects on body weight from start to end of treatment after the addition or substitution with finerenone.
(Additive) treatment effects finerenone on eGFR | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  (Additive) treatment effects on eGFR from start to end of treatment after the addition or substitution with finerenone.
(Additive) treatment effects finerenone on fasting plasma glucose | Will be assessed within 6 months and reported within 1 year after conclusion of the study.
  (Additive) treatment effects on fasting plasma glucose from start to end of treatment after the addition or substitution with finerenone.

CONTACTS AND LOCATIONS:
Overall Officials: Hiddo Lambers Heerspink, Principal Investigator — University Medical Center Groningen
Locations (1):
- ZorgGroep Twente, Almelo, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Yes